CLINICAL TRIAL: NCT07371689
Title: ANAKINRA IN THE TREATMENT OF PEDIATRIC ACUTE MYOCARDITIS
Acronym: ANAPEM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP230825; 2025-521478-32-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: PEDIATRIC ACUTE MYOCARDITIS
Keywords: Myocarditis; Anakinra; Anti-IL1; Inflammation; Pediatric
MeSH Terms: conditions — Myocarditis; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: This is a superiority, national multicentre phase III double-blind randomized placebo-controlled trial to demonstrate the efficacy of Anakinra vs placebo as an add-on curative treatment on top of standard of care of acute myocarditis in children.
  Diagnosis of myocarditis is confirmed, in addition to troponin T rise (*1.5 Normal range), by an echocardiogram performed during the first 24H of suspicion.
  Patients will be randomized to receive Anakinra 4mg/Kg (maximum 100 mg) or placebo subcutaneously once a day for 7 days, in addition to standard care: ACE and/or Beta-blocker.
  Randomization 1:1 will be conducted centrally with the use of an Interactive WEB Randomisation system (IWRS).
  Patients who have failed at 3 days of treatment will be treated at the clinicians' discretion and can receive anakinra.
  Discharge will be left to the physician decision, based on the normalization of systolic function and troponin T, and lack of complication defined by heart failure, ventricular ta
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anakinra (Experimental): Anakinra, KINERET, solution for injection in pre-filled syringe. Posology for clinical trial: 4 mg/Kg (maximum 100 mg) once daily subcutaneously for 7 days.
  Interventions: Drug: Anakinra, KINERET®
- Placebo (Placebo Comparator): Placebo of Anakinra, solution of NaCl 0.9% Posology for clinical trial: 4 mg/Kg (maximum 100 mg) once daily subcutaneously for 7 days.
  Interventions: Drug: Anakinra, KINERET®

INTERVENTIONS:
Drug: Anakinra, KINERET® — Patients will be randomized to receive Anakinra 4mg/Kg (maximum 100 mg) subcutaneously once a day for 7 days

SUMMARY:
Double blind RCT aiming to compare the efficacy of Anakinra vs placebo, on top of the standard of care, on restoration of myocardial function at 3 days following treatment initiation, in children admitted for acute myocarditis in intensive care units.

DETAILED DESCRIPTION:
Activation of the inflammasome is increasingly recognized in the pathogenesis of acute myocarditis. We hypothesize that by blocking inflammasome using anakinra, we interfere with the key mechanism driving myocardial inflammation and fibrosis, allowing for restauration of myocardial function compared to standard of care alone. Children from ≥ 3 months to < 18 years of age hospitalized in the Intensive Care Unit for acute myocarditis defined as a reduced left ventricle ejection fraction below 50% and troponin T rise (>1.5x normal range) will be randomized to either receive SC Anakinra or Placebo in addition to standard of care treatment. Primary endpoint: Proportion of children with recovered left ventricle ejection fraction (LVEF ≥ 50%) measured by echocardiography at 3 days after treatment initiation.

Secondary endpoints:

1. Proportion of children with recovered left ventricle ejection fraction (LVEF

   ≥ 50%) measured by echocardiography at 7 and 28 days after treatment initiation. Patients who die or undergo heart transplant within the first 7 and 28 days after treatment initiation respectively will be considered as a failure (i.e, LVEF < 50%). Patients who still require ECMO at 7 and 28 days after treatment initiation respectively will also be considered as failure (i.e., LVEF < 50%).
2. Time to recovery of normal left ventricular ejection fraction (LVEF ≥ 50%) within the first 3 days after treatment initiation
3. Proportion of children requiring ECMO within the first 3 days after treatment initiation
4. Proportion of children who undergo heart transplant within 6 months after treatment initiation
5. Time to all-cause death within 6 months after treatment initiation
6. Time to cardiovascular-related death within 6 months after treatment initiation
7. Proportion of children with drug-related side effects (hypersensitivity, neutropenia, drug-related liver enzymes elevation…)
8. a- NT proBNP at inclusion and at 24 hours, 48 hours, 72 hours following treatment initiation - Troponin T at inclusion and at 24 hours, 48 hours, 72 hours following treatment initiation - Proportion of children with ventricular tachycardia assessed by EKG at inclusion and at 24 hours, 48 hours, 72 hours following treatment initiation - b - NT proBNP at 7 days following treatment initiation - Troponin T at 7 days following treatment initiation - Proportion of children with ventricular tachycardia assessed by EKG at 7 days following treatment initiation - Proportion of children with fibrosis on cardiac MRI according to modified Lake Louise criteria at 6 months following treatment initiation - Proportion of children with dilated cardiomyopathy on cardiac echocardiography (Left ventricular end diastolic diameter ˃ 2 SD with altered systolic function <50%) at 3 and 6 months following treatment initiation - Proportion of children with ventricular arrhythmia at 6 months following treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Children from ≥ 3 months to < 18 years of age
* Hospitalized in the Intensive Care Unit (ICU) for acute myocarditis defined as : - a reduced left ventricle ejection fraction below 50% and - troponin T rise (>1.5x normal range), Signed informed consent by legal representative and patient according to the legislation.

Exclusion Criteria:

* Children weighing less than 5 Kgs
* Known anterior cardiomyopathy or operated cardiopathy
* Neutropenia (< 1,5 × 10^9 /L).
* Known hypersensitivity to Anakinra or any of its excipients (citric acid anhydrous, sodium chloride, disodium EDTA dihydrate, polysorbate 80, E. coli derived proteins)
* Administration of a live vaccine in the 4 weeks prior to inclusion
* Hepatitis B infection, defined as positive HBsAg and/or detectable HBV DNA (PCR). Patients with increased risk of Tuberculosis (TB) infection
* Recent tuberculosis infection or with active TB

  * Close contact with a patient with TB
  * Patients recently arrived less than 3 months from a country with high prevalence of TB
  * A chest radiograph suggestive of TB
* Patients with overt concomitant bacterial infection
* Patients previously treated with another biotherapy
* Patients with any type of immunodeficiency or cancer
* Anti TNF-α within the past 14 days
* Malignancy or history of malignancy or any comorbidity limiting survival or conditions predicting inability to complete the study Ongoing or recent use of any other medication Known inhibitors/inducers of cytochrome P450
* Pregnancy or breastfeeding
* No affiliation to the Social Security
* Current enrollment in another clinical trial
* Inability of the legal representative (and the patient, when applicable) to understand the national language (French)

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of children with recovered left ventricle ejection fraction ≥ 50% measured by echocardiography at 3 days after treatment initiation. | 3 days
  Main objective: To compare the efficacy of Anakinra vs placebo, on top of the standard of care, on restoration of myocardial function at 3 days following treatment initiation, in children admitted for acute myocarditis in intensive care units. Primary endpoint: Proportion of children with recovered left ventricle ejection fraction (LVEF ≥ 50%) measured by echocardiography at 3 days after treatment initiation. Patients who die within the first 3 days after treatment initiation or patients who still require ECMO at 3 days after treatment initiation will be considered as a failure.

SECONDARY OUTCOMES:
Proportion of children with recovered left ventricle ejection fraction ≥ 50% measured by echocardiography at 7 and 28 days after treatment initiation. Patients who die or undergo heart transplant within the first 7 and 28 days after treatment initiation | 7 and 28 days
Time to recovery of normal left ventricular ejection fraction (LVEF ≥ 50%) within the first 3 days after treatment initiation | 3 days
Proportion of children requiring ECMO within the first 3 days after treatment initiation | 3 days
Proportion of children who undergo heart transplant within 6 months after treatment initiation | 6 months
Time to all-cause death within 6 months after treatment initiation | 6 months
Time to cardiovascular-related death within 6 months after treatment initiation | 6 months
Proportion of children with drug-related side effects (hypersensitivity, neutropenia, drug-related liver enzymes elevation…) | 6 months
following treatment initiation-TroponinT at inclusion and at24 hours,48 hours,72 hours following treatment initiation-Proportion of children with ventricular tachycardia assessed by EKG at inclusion and at 24hours,48hours,72hours following treatment init | 24,48,72 hours
NTproBNP at7days, Troponin T at7days,Proportion of children with ventricular tachycardia assessed by EKG at7days, Proportion of children with fibros on cardiac MRI at6months,Proportion of children with dilated cardiomyopathy,with ventricular arrhythmia | 7 days - 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bicêtre Hospital - APHP, Pediatric intensive care unit, Le Kremlin-Bicêtre, France, France

IPD SHARING:
Plan to Share IPD: No